CLINICAL TRIAL: NCT02502552
Title: Study of Anti-glycan Antibodies Stability in Saint-Etienne IBD Cohort - A Monocentric Study
Brief Title: Study of Anti-glycan Antibodies Stability in Saint-Etienne IBD Cohort
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1308018
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease; anti-glycan antibodies; antibodies stability; mucosal healing; predictive markers
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimen in IBD cohort of 195 patients followed in Saint-Etienne Hospital
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inflammatory Bowel Disease: Inflammatory Bowel Disease patients followed in Saint-Etienne Hospital since 3 years or more. Blood specimen 3 years after a first blood specimen
  Interventions: Other: blood specimen

INTERVENTIONS:
Other: blood specimen — blood specimen

SUMMARY:
Prognostic factors in Inflammatory Bowel Diseases (IBD) are currently mainly based on clinical factors (disease extension, perianal involvement, need for surgery, use of immunomodulators…). All of immunological markers (or serological) of IBD have a diagnostic role in indeterminate colitis (ulcerative colitis vs crohn's disease) but they never have been considered as predictors of IBD course in adults. Among the most used, anti-neutrophil cytoplasm antibodies (ANCA) and Anti-Saccaromyces cerevisiae antibodies (ASCA) allow the distinction between ulcerative colitis (ANCA+/ASCA-) and Crohn's disease (ANCA-/ASCA+), and their combined use has a sensitivity and a specificity of about 85%. However, 10 other antibodies have been identified and recently evaluated individually in IBD and especially in pediatric Crohn's disease: anti-ompC, anti-I2, anti-flagellins, anti-glycan (anti-laminaribioside carbohydrate antibodies (ALCA), anti-mannobioside carbohydrate antibodies (AMCA), anti-chitobioside carbohydrate antibody (ACCA), anti-chitin and anti-laminarin), anti-goblet cells and anti-C.albicans specific mannans antibodies. These complementary tests improve the reliability of the diagnosis. In a previous cross-sectional work on a cohort of 195 IBD patients, the investigator showed a prognostic role of some of anti-glycan Abs and especially a correlation with a pejorative form of the disease both in Crohn's disease than in Ulcerative Colitis (UC) and a prediction of corticodependency in IBD.

DETAILED DESCRIPTION:
There is few data on the stability of these antibodies, most of the studies are cross-sectional. There are conflicting results among scarce longitudinal data. One study reported a negativation of anti-glycan antibodies in some cases but not of ASCA or ANCA.

On the cohort of 195 patients included in the first study, the investigator would like to assess at 3 years the immunological profiles of these patients and thus to compare them. In case of modification of the serological status for some antibodies, the search for associated factors (clinical, biological or therapeutic) will be performed. In case of sero-negativation of anti-glycan antibodies, this could be linked with a decrease or a normalization of the increased intestinal permeability in IBD. Indeed, in this subgroup of patients, we will test this hypothesis by analyzing intestinal permeability in anti-glycan positive group on the 2 samples and in the group with a sero-negativation on the second sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in previous study (AOL 2010) and followed in our department, accepting blood sampling and stool analysis
* Written consent of the patient

Exclusion Criteria:

* Patient who decline to participate to the study
* Patient in the incapacity to give consent
* Patient deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ulcerative colitis and Crohn's disease patient followed in Saint-Etienne Hospital since 3 years or more
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
immunological status | 3 years after first evaluation
  Immunological status is defined by anti-glycan antibodies (ACCA, ALCA, AMCA, anti-chitin and anti-laminarin), ASCA and ANCA.
  Antibody will be positive if level is found higher than the threshold defined by the laboratory (technical threshold).
  An antibody will be defined as stable if its status remains positive during 3 years(above the detection limit given by the reference laboratory) or negative during 3 years (below the detection limit given by the reference laboratory). Conversely, the lack of stability during 3 years will be defined as the transition from a positive to a negative status or inversely.

SECONDARY OUTCOMES:
clinical remission | 3 years after first evaluation
  Comparison of clinical remission between patients with a change in their immunological status and patients with stable status.
  A patient is in clinical remission if:
  1. Crohn's disease activity index (CDAI) score is lower than 150 for Crohn's disease
  2. Lichtiger score is < 4 for Ulcerative Colitis
anti-Tumor Necrosis Factor (TNF) therapeutic response | 3 years after first evaluation
  Comparison of anti-TNF (Tumor Necrosis Factor) therapeutic response between patients with a change in their immunological status and patients with stable status.
  A patient is considered as anti-TNF responder if there is a clinical remission without therapeutic change in the medical history of the patient
Mucosal healing | 3 years after first evaluation
  Comparison of mucosal healing between patients with a change in their immunological status and patients with stable status.
  A patient will be considered in mucosal healing if:
  1. C-reactive Protein (CRP) < 5mg/L and fecal calprotectin <250 µg/g
  2. Fecal calprotectin <150 µg/g in Ulcerative colitis
Intestinal permeability | 3 years after first evaluation
  Comparison of intestinal permeability between patients with a change in their immunological status and patients with stable status.
  4. Normalization of intestinal permeability will be defined if lipopolysaccharide (LPS) or anti-LPS Antibodies (IgG) level measured by LAL or ELISA is significantly reduced between the two samples. As there is no pre-defined threshold for LPS and anti-LPS Antibodies level in normalization of intestinal permeability, we will calculate a delta (level before - level at 3 years) for each patient and each parameter. We will analyze the average delta with the stability or not of immunological status.
surgical resection | 3 years after first evaluation
  Comparison of number of surgical resection between patients with a change in their immunological status and patients with stable status.
  5. Surgical resection may be a colonic or small bowel resection surgery for CD patients or colectomy for UC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Roblin, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France